CLINICAL TRIAL: NCT05240963
Title: Patient Specific PEEK Implants for Immediate Restoration of Temporal Fossa After Maxillary Reconstruction With Temporalis Muscle Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Ali, Associate Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS-19715
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Temporal Hollowing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK implant (Experimental): Temporal PEEK implant to prevent temporal hollowing after temporalis muscle transfer
  Interventions: Procedure: Temporal PEEK implant

INTERVENTIONS:
Procedure: Temporal PEEK implant — Temporal PEEK implant to reconstruct temporal fossa after temporalis muscle transfer

SUMMARY:
Study conducted on patients with major maxillary defects indicating the need of reconstruction with full temporalis muscle flap; or any lesion indicating major maxillary resection and immediate reconstruction with total temporalis muscle flap.

For each patient, a patient specific PEEK implant was fabricated, the temporalis muscle was exposed, elevated, and transferred to the maxilla, finally PEEK implants were fixed in place to prevent temporal hollowing.

DETAILED DESCRIPTION:
Study conducted on patients with major maxillary defects indicating the need of reconstruction with full temporalis muscle flap; or any lesion indicating major maxillary resection and immediate reconstruction with total temporalis muscle flap.

For each patient, a patient specific PEEK implant was fabricated, the temporalis muscle was exposed, elevated, and transferred to the maxilla, finally PEEK implants were fixed in place to prevent temporal hollowing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with major maxillary defects indicating the need of reconstruction with full temporalis muscle flap; or any lesion indicating major maxillary resection and immediate reconstruction with total temporalis muscle flap.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
patient's satisfaction | 3 weeks postoperative
  patient's satisfaction using five points Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali S, Abdel Aziz O, Ahmed M. Patient-specific PEEK implants for immediate restoration of temporal fossa after maxillary reconstruction with temporalis muscle flap. Maxillofac Plast Reconstr Surg. 2022 May 7;44(1):20. doi: 10.1186/s40902-022-00348-4. PMID 35524015